CLINICAL TRIAL: NCT07037979
Title: Correlation of Sarcopenia and Peripheral Artery Disease With Chronic Limb Threatening Ischemia
Brief Title: Sarcopenia and Peripheral Artery Disease With Chronic Limb Threatening Ischemia
Acronym: SAC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Hospital director, Fudan University
Other Study IDs: 2025ZW02
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia; Peripheral Arterial Disease; Chronic Limb Threatening Ischemia
MeSH Terms: conditions — Sarcopenia; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patiets with peripheral artery disease
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — non-applicable

SUMMARY:
To evaluate the correlation of Sarcopenia Parameters and Peripheral Artery Disease with chronic limb threatening ischaemia.

DETAILED DESCRIPTION:
Prior researches indicated a relatively high prevalence of sarcopenia among patients of Peripheral Artery Disease. However, the relationship between sarcopenia and progression of Peripheral Artery Disease with chronic limb threatening ischaemia remained poorly understood. Thus, this cohort study aimed to evaluate the correlation of Sarcopenia Parameters, such as psoas muscle area (PMA) and total abdominal muscle area (TAMA) at the L3 vertebral level, measured by computed tomography (CT), and progression of Peripheral Artery Disease with chronic limb threatening ischaemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Peripheral Artery Disease, including intermittent claudication and Chronic Limb Threatening Ischemia;
* Patients with Rutherford grade 2-6 between Jan.1 2023 and Dec.31 2024;
* Patients at age 18-80;
* Patients underwent an in-hospital routine enhanced whole abdomen to lower extremities CT scan;
* Patients able to complete the clinical follow-up for 3 months.

Exclusion Criteria:

* Poor CT quality or incomplete images;
* Incomplete clinical data;
* In-hospital mortality during Jan.1 2023 and Dec.31 2024.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: patients of Peripheral Artery Disease
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
psoas muscle area (PMA) [measured by computed tomography (CT)] | 2023.1.1～2024.12.31
  psoas muscle area (PMA) (square centimeters) was regarded as a kind of typical sarcopenia parameters, measured by computed tomography (CT) at the L3 vertebral level
total abdominal muscle area (TAMA) measured by computed tomography (CT) | 2023.1.1～2024.12.31
  total abdominal muscle area (TAMA) (square centimeters) was regarded as a kind of typical sarcopenia parameters, measured by computed tomography (CT) at the L3 vertebral level

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided